CLINICAL TRIAL: NCT06761989
Title: Effect of Single-Shot Intrathecal Morphine Injection Versus Continuous Wound Infiltration on Postoperative Pain After Pancreaticoduodenectomy: a Prospective, Open-Label, Randomized Controlled, Non-Inferiority Trial
Brief Title: Intrathecal Morphine Injection Versus Continuous Wound Infiltration After Pancreaticoduodenectomy
Acronym: ITM_PPPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hojin Lee, MD, PhD, Associated Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-2411-020-1585
Record Dates: First submitted 2024-12-30; First posted 2025-01-07 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Pain Management; Pain, Postoperative
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Stratify patients who receive preoperative chemotherapy and those who do not in a 1:3 ratio, so that 26 and 78 patients are assigned to each stratum out of a total of 104 patients. Then, within each stratum, block randomization is performed, with blocks of size 4 containing two intrathecal morphine and two wound infiltration groups, and blocks of size 6 containing three intrathecal morphine and three wound infiltration groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intrathecal morphine injection (Experimental): A single dose of intrathecal morphine is administered prior to induction of general anesthesia. Other postoperative pain management follows the institution's protocol including intravenous patient controlled analgesia.
  Interventions: Drug: Intrathecal morphine injection
- Continuous wound infiltration (Active Comparator): A catheter is inserted at preperitoneal space at the end of surgery and ropivacaine is continuously infused until postoperative day 3. Other postoperative pain management follows the institution's protocol including intravenous patient controlled analgesia.
  Interventions: Device: Continuous wound infiltration

INTERVENTIONS:
Drug: Intrathecal morphine injection — A single dose of intrathecal morphine is administered prior to induction of general anesthesia. The patient is placed in the lateral decubitus position on the bed and a 25 guage quincke spinal needle is inserted intrathecally at the L4/5 median or paramedian approach to administer 0.2 mg of morphine.
  Arms: Intrathecal morphine injection
Device: Continuous wound infiltration — Prior to closure of the abdominal wall, a catheter is placed in the preperitoneal space lateral to the surgical incision through the tunneler. The catheter is connected to a prepared infusion pump (275 ml of 0.5% ropivacaine, 4 ml/hr/catheter), and the remaining catheter protruding from the abdomen is secured with a catheterization dressing. The preperitoneal catheter is removed in the afternoon of postoperative day 3.
  Arms: Continuous wound infiltration

SUMMARY:
This is a prospective randomized open-label noninferiority trial that compares intrathecal morphine injection and continuous wound infiltration after open pancreaticoduodenectomy.

DETAILED DESCRIPTION:
Open pancreaticoduodenectomy causes severe postoperative pain due to the relatively large incision and tissue damage compared to other abdominal surgeries. Current Enhanced Recovery After Surgery (ERAS) guidelines recommend continuous wound infiltration for pancreaticoduodenectomy as an effective analgesic modality along with thoracic epidural analgesia. However, continuous wound infiltration is effective for somatic pain in the abdominal wall but not for visceral pain from the incision of internal organs. It also requires the placement of a catheter for several days after surgery, which can be inconvenient for patients.

Intrathecal morphine injection has been recommended as an effective analgesic method for abdominal surgery because they provide potent, long-lasting analgesia with a single injection and can provide equivalent analgesia with a much smaller dose compared to intravenous or oral morphine. Several previous studies have reported on the analgesic efficacy of a single intrathecal morphine injection including pancreaticoduodenectomy. However, no studies have compared a single intrathecal morphine injection with continuous wound infiltration for pancreaticoduodenectomy. To date, studies comparing the two methods of analgesia have only been reported in cesarean section and donor hepatectomy, and these studies either found no significant difference between the two methods of analgesia or reported that intrathecal morphine injection provided better analgesia in early postoperative period.

Therefore, the investigators will examine the effect of single intrathecal morphine injection for postoperative pain control in patients undergoing open pancreaticoduodenectomy to improve postoperative pain management and to explore its potential as one of the effective analgesic methods in ERAS protocol. To this end, the investigators will test non-inferiority between intrathecal morphine injection and continuous wound infiltration.

ELIGIBILITY:
Inclusion Criteria:

* Adults 19 years of age or older
* Scheduled for elective open pancreaticoduodenectomy or pylorus preseriving pancreaticoduodenectomy
* Disease of periampullary lesions
* Perfromance status assessed with ECOG score is 0 or 1 at the time of enrollment
* Able to provide written informed consent to participate in the study, understand the procedures of this study, and complete patient-reported questionnaires
* American Society of Anesthesiologists physical status I to III

Exclusion Criteria:

* Hypersensitivity to medications used for pain control (fentanyl, ropivacaine, morphine, acetaminophen, NSAIDs)
* Cognitive impairment that affects using patient-controlled analgesia device or answering patient-reported questionnaires
* Infection or anatomical abnormalities of the abdominal wall and skin that preclude catheterization for continuous wound infiltration
* Contraindicated for intrathecal injection due to any coagulation disorder or continued use of anticoagulants
* Have a major medical or psychiatric illness that would affect response to treatment
* History of chronic pain, or chronic use of analgesics or psychiatric medications
* Have severe liver or kidney disease
* Anyone who are not appropriate for the study in the opinion of the investigators

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-07 (Estimated)

PRIMARY OUTCOMES:
Mean pain intensity on cough assessed by K-DVRPS at 24, 48, and 72 hours from the end of anesthesia | Postoperative days 1 to 3
  The K-DVPRS (Korean version of Defense and Veterans Pain Rating Scale), ranging from 0 to 10, is used to assess postoperative pain on cough at 24, 48, and 72 hours after the end of anesthesia. The mean K-DVPRS pain score for 3 time points is compared between two groups.

SECONDARY OUTCOMES:
Mean pain intensity at rest assessed by K-DVRPS at 24, 48, and 72 hours from the end of anesthesia | Postoperative days 1 to 3
  The K-DVPRS is used to assess postoperative pain at rest at 24, 48, and 72 hours after the end of anesthesia. The mean K-DVPRS pain score for 3 time points is compared between two groups.
Pain intensity at rest and on cough assessed at 2, 24, 48, and 72 hours from end of anesthesia | Postoperative days 0 to 3
  The K-DVPRS is used to assess postoperative pain at rest and on cough at 2, 24, 48, and 72 hours after the end of anesthesia, respectively.
Cumulative dose of opioid use at 6, 12, 24, 48, and 72 hours after end of anesthesia | Postoperative days 0 to 3
  The cumulative fentanyl equivalent dose used at 6, 12, 24, 48, and 72 hours after the end of anesthesia is assessed.
Quality of recovery at 24, 48, and 72 hours from the end of anesthesia | Postoperative days 1 to 3
  Quality of recovery is assessed with the Korean version of the EQ-5D-5L at 24, 48, and 72 hours after the end of anesthesia.
Postoperative complications | Within 1 week after surgery
  Postoperative complications are assessed with the comprehensive complication index.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided